CLINICAL TRIAL: NCT03460197
Title: Capillarity Versus Wet Technique. Comparison Between Two Methods of Tissue Acquisition Guided by Endoscopic Ultrasound.
Brief Title: Comparison Between Two Tissue Acquisition Techniques by Endoscopic Ultrasound. (EUS)
Acronym: EUS
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Dulce Maria Rascon Martinez, MD Clinical Researcher., Instituto Mexicano del Seguro Social
Other Study IDs: R-2016-3601-190
Record Dates: First submitted 2018-01-12; First posted 2018-03-09 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Digestive Cancer
Keywords: Capillary technique; Wet technique; Endoscopic Ultrasound-Guided Fine-Needle Aspiration
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsies of suspicious digestive tumors obtained by endoscopic -ultrasound. Cellularity and sample quality will be documented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic Ultrasound-Guided Fine-Needle Aspiration — Patients will be submitted to both techniques of tissue acquisition in the same procedure of endoscopic ultrasound. Capillarity technique, requires not remove the stiletto from the needle until the punctures are done for the biopsy sampling. Wet suction technique, requires saline solution to replace the air column. Samplings will be placed in two different jars, where Jar 1 corresponds to Capillarity Technique sampling and Jar 2 to Wet Technique. Once the sampling preparation is concluded will be send to the Pathology Department to be subsequently blindly analyzed by two independent pathologists, that means they would not be aware of the tissue acquisition method used in each of the microscopic slides to analyze.

SUMMARY:
There are various techniques to obtain tissue samples by using fine needle guided by endoscopic ultrasound (EUS). These techniques attempt to obtain the most adequate material with the best quantity and quality for analysis. Currently studies that compare the results concerning capillary technique versus wet technique are not available. In this sense, the authors consider necessary to explore both techniques documenting the results that can define which could be the best method so that it can routinely be used in cases of digestive neoplasia.

DETAILED DESCRIPTION:
The aim of the study will be compare both techniques guided by endoscopic ultrasound (Capillarity versus Wet) and identify which obtains the best sample quality for histopathology analysis as tissue acquisition method in patients diagnosed with tumors of pancreas, biliary tract, liver or lymph nodes.

The researchers are planning a prospective, pilot study in 30 subjects. All patients will be submitted to both techniques of tissue acquisition (capillarity versus wet) in the same procedure of endoscopic ultrasound. Obtained samples for histopathology analysis will be submitted to a blind examination by two different pathologists.

ELIGIBILITY:
Inclusion Criteria:

* Low or moderate suspicious of malignancy lesion in pancreas, liver or metastatic lymph nodes
* Initial diagnosis according to the characterization by endoscopic ultrasound

Exclusion Criteria:

* Bleeding
* Complications during biopsy procedure
* Needed to use procedures other than those contemplated in the study.
* Patients who not require endoscopic ultrasound evaluation
* Patients who not accept the procedures of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Referred to the Endoscopy Department from their corresponding basic health care units within the Mexican Social Security System
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
The classification of Papanicolaou was used for the terminology in pancreatobiliary cytological evaluation of biopsy samples. | 4 months once the study has begun
  I.- Non-diagnostic: Specimen does not provide information about whether the lesion is cystic or solid.
  II.- Negative (for malignancy): Specimen has adequate cellularity and / or extracellular material that defines a lesion that is identified by image.
  III.- Atypical: There are cells with architectural, nuclear or cytoplasmic that are not consistent with reactive changes. However, these findings are not conclusive to diagnose malignancy or suspected of malignancy.
  IV.- Neoplastic: benign and others. Neoplasic benign: Sample has elements of benign neoplasm. Neoplastic others: May be is a premalignant lesion like low-level dysplasia, intermediate or high grade dysplasia or a low grade neoplasm with malignant behavior.
  V.- Suspected of malignancy: Cytological characteristics support the Diagnosis of malignancy but quantitatively or qualitatively is not enough to confirm it.
  VI.- Positive / malignant: Cytological changes are unequivocal of malignancy.

CONTACTS AND LOCATIONS:
Overall Officials: Dulce M. Rascon, M.D, Study Director — Instituto Mexicano del Seguro Social; Alejandro Membrillo, Endoscopist, Principal Investigator — Instituto Mexicano del Seguro Social; Luis F. Palacio, Endoscopist, Study Chair — Instituto Mexicano del Seguro Social; Luz M. Gomez, Pathologist, Study Chair — Instituto Mexicano del Seguro Social; Yelitzia A. Valverde, Pathologist, Study Chair — Instituto Mexicano del Seguro Social
Locations (1):
- Centro Medico Nacional Siglo XXI. UMAE Hospital de Especialidades, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
This is a pilot study. It means a few patients will be included. We are not subjecting the participants to a higher risk than the endoscopic ultrasound itself and the procedures performed here are usual. The authors will only document the experience.

REFERENCES:
- [Background] Attam R, Arain MA, Bloechl SJ, Trikudanathan G, Munigala S, Bakman Y, Singh M, Wallace T, Henderson JB, Catalano MF, Guda NM. "Wet suction technique (WEST)": a novel way to enhance the quality of EUS-FNA aspirate. Results of a prospective, single-blind, randomized, controlled trial using a 22-gauge needle for EUS-FNA of solid lesions. Gastrointest Endosc. 2015;81(6):1401-7. doi: 10.1016/j.gie.2014.11.023. Epub 2015 Feb 27. PMID 25733127
- [Background] Polkowski M, Jenssen C, Kaye P, Carrara S, Deprez P, Gines A, Fernandez-Esparrach G, Eisendrath P, Aithal GP, Arcidiacono P, Barthet M, Bastos P, Fornelli A, Napoleon B, Iglesias-Garcia J, Seicean A, Larghi A, Hassan C, van Hooft JE, Dumonceau JM. Technical aspects of endoscopic ultrasound (EUS)-guided sampling in gastroenterology: European Society of Gastrointestinal Endoscopy (ESGE) Technical Guideline - March 2017. Endoscopy. 2017 Oct;49(10):989-1006. doi: 10.1055/s-0043-119219. Epub 2017 Sep 12. PMID 28898917
- [Background] Lakhtakia S. Complications of diagnostic and therapeutic Endoscopic Ultrasound. Best Pract Res Clin Gastroenterol. 2016 Oct;30(5):807-823. doi: 10.1016/j.bpg.2016.10.008. Epub 2016 Oct 28. PMID 27931638
- [Background] Wiersema MJ, Kochman ML, Cramer HM, Tao LC, Wiersema LM. Endosonography-guided real-time fine-needle aspiration biopsy. Gastrointest Endosc. 1994 Nov-Dec;40(6):700-7. PMID 7859968
- [Background] Hedenstrom P, Demir A, Khodakaram K, Nilsson O, Sadik R. EUS-guided reverse bevel fine-needle biopsy sampling and open tip fine-needle aspiration in solid pancreatic lesions - a prospective, comparative study. Scand J Gastroenterol. 2018 Feb;53(2):231-237. doi: 10.1080/00365521.2017.1421704. Epub 2018 Jan 4. PMID 29301477
- [Background] Ang TL, Kwek ABE, Wang LM. Diagnostic Endoscopic Ultrasound: Technique, Current Status and Future Directions. Gut Liver. 2018 Sep 15;12(5):483-496. doi: 10.5009/gnl17348. PMID 29291601
- [Background] Wani S, Muthusamy VR, Komanduri S. EUS-guided tissue acquisition: an evidence-based approach (with videos). Gastrointest Endosc. 2014 Dec;80(6):939-59.e7. doi: 10.1016/j.gie.2014.07.066. No abstract available. PMID 25434654
- [Background] Varadarajulu S, Hasan MK, Bang JY, Hebert-Magee S, Hawes RH. Endoscopic ultrasound-guided tissue acquisition. Dig Endosc. 2014 Jan;26 Suppl 1:62-9. doi: 10.1111/den.12146. Epub 2013 Aug 28. PMID 24033879
- [Background] Jani BS, Rzouq F, Saligram S, Lim D, Rastogi A, Bonino J, Olyaee M. Endoscopic Ultrasound-Guided Fine-Needle Aspiration of Pancreatic Lesions: A Systematic Review of Technical and Procedural Variables. N Am J Med Sci. 2016 Jan;8(1):1-11. doi: 10.4103/1947-2714.175185. PMID 27011940
- [Background] Wang J, Wu X, Yin P, Guo Q, Hou W, Li Y, Wang Y, Cheng B. Comparing endoscopic ultrasound (EUS)-guided fine needle aspiration (FNA) versus fine needle biopsy (FNB) in the diagnosis of solid lesions: study protocol for a randomized controlled trial. Trials. 2016 Apr 12;17:198. doi: 10.1186/s13063-016-1316-2. PMID 27071386
- [Background] Iwashita T, Nakai Y, Samarasena JB, Park DH, Zhang Z, Gu M, Lee JG, Chang KJ. High single-pass diagnostic yield of a new 25-gauge core biopsy needle for EUS-guided FNA biopsy in solid pancreatic lesions. Gastrointest Endosc. 2013 Jun;77(6):909-15. doi: 10.1016/j.gie.2013.01.001. Epub 2013 Feb 20. PMID 23433596
- [Background] Bang JY, Hawes RH, Varadarajulu S. EUS-guided tissue acquisition: things are not always what they seem. Gastrointest Endosc. 2015 May;81(5):1300-1. doi: 10.1016/j.gie.2014.12.044. No abstract available. PMID 25864902
- [Background] Vilmann P, Seicean A, Saftoiu A. Tips to overcome technical challenges in EUS-guided tissue acquisition. Gastrointest Endosc Clin N Am. 2014 Jan;24(1):109-24. doi: 10.1016/j.giec.2013.08.009. PMID 24215763
- [Background] Shah JN, Muthusamy VR. Minimizing complications of endoscopic ultrasound and EUS-guided fine needle aspiration. Gastrointest Endosc Clin N Am. 2007 Jan;17(1):129-43, vii-viii. doi: 10.1016/j.giec.2006.10.002. PMID 17397780
- [Background] Yamao K, Ohashi K, Mizutani S, Furukawa T, Watanabe Y, Nakamura T, Suzuki T, Takeda K. Endoscopic ultrasound-guided fine-needle aspiration (EUS-FNA) for the diagnosis of digestive diseases. Endoscopy. 1998 Aug;30 Suppl 1:A176-8. doi: 10.1055/s-2007-1001513. No abstract available. PMID 9765119
- [Background] Puri R, Vilmann P, Saftoiu A, Skov BG, Linnemann D, Hassan H, Garcia ES, Gorunescu F. Randomized controlled trial of endoscopic ultrasound-guided fine-needle sampling with or without suction for better cytological diagnosis. Scand J Gastroenterol. 2009;44(4):499-504. doi: 10.1080/00365520802647392. PMID 19117242
- [Background] Panic N, Larghi A. Techniques for endoscopic ultrasound-guided fine-needle biopsy. Gastrointest Endosc Clin N Am. 2014 Jan;24(1):83-107. doi: 10.1016/j.giec.2013.08.010. PMID 24215762
- [Background] Yamao K, Bhatia V, Mizuno N, Sawaki A, Shimizu Y, Irisawa A. Interventional endoscopic ultrasonography. J Gastroenterol Hepatol. 2009 Apr;24(4):509-19. doi: 10.1111/j.1440-1746.2009.05783.x. PMID 19220671
- [Background] Wee E, Lakhtakia S, Gupta R, Sekaran A, Kalapala R, Monga A, Arjunan S, Reddy DN. Endoscopic ultrasound guided fine-needle aspiration of lymph nodes and solid masses: factors influencing the cellularity and adequacy of the aspirate. J Clin Gastroenterol. 2012 Jul;46(6):487-93. doi: 10.1097/MCG.0b013e31824432cb. PMID 22688144
- [Background] Hollerbach S, Juergensen C, Hocke M, Freund U, Wellmann A, Burmester E. [EUS-FNA: how to improve biopsy results? An evidence based review]. Z Gastroenterol. 2014 Sep;52(9):1081-92. doi: 10.1055/s-0034-1385133. Epub 2014 Sep 8. German. PMID 25198088
- [Background] Paquin SC, Sahai AV. Techniques for EUS-guided FNA cytology. Gastrointest Endosc Clin N Am. 2014 Jan;24(1):71-81. doi: 10.1016/j.giec.2013.08.007. PMID 24215761